CLINICAL TRIAL: NCT01084148
Title: Long-term Efficacy and Safety of V0034 CR 01B Cream in Patients With Moderate-to-severe Uremic Xerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orfagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V00034 CR 308 ORF
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Uremic Xerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- V0034CR01B (Experimental): cream
  Interventions: Drug: V0034CR01B
- V0034 CR 01B vehicle (Placebo Comparator): cream
  Interventions: Drug: V0034CR01B vehicle

INTERVENTIONS:
Drug: V0034CR01B
  Arms: V0034CR01B
Drug: V0034CR01B vehicle
  Arms: V0034 CR 01B vehicle

SUMMARY:
Primary objective:

To demonstrate the long-term efficacy (response to treatment during initial therapy, time to relapse without treatment, durability and lesional recurrence during maintenance therapy) of V0034 CR 01B cream on uraemic xerosis in the real-life setting.

Secondary objectives:

1. To assess the local tolerance of V0034 CR 01B after long-term use
2. To assess the patient benefit and acceptability of V0034 CR 01B

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, of at least 18 years of age
2. Women of childbearing potential having a reliable contraceptive method
3. Patients undergoing maintenance renal dialysis (MRD), i.e. either haemodialysis or peritoneal dialysis, due to chronic renal failure
4. Patients whose xerosis is related to their renal insufficiency status (uraemic xerosis)
5. Patients suffering from xerosis with a severity score of at least two, on at least one of the five tests areas (right lower leg, left lower leg, forearm with no arterio-venous shunt, chest, dorsum of the neck)

Exclusion Criteria:

1. Patients under 18 years of age
2. Women with childbearing potential having a positive pregnancy test at baseline
3. Patients undergoing renal dialysis for another reason than chronic renal insufficiency
4. Patients whose xerosis is due to another reason than their MRD status
5. Patients suffering from mild xerosis (i.e. score less than two on all the xerotic test areas)
6. Patients with a known history of allergy to one of the ingredients contained in the test product
7. Patients with an intercurrent condition which may interfere with a good conduct or the study parameters of the study
8. Patients treated with any other emollient/moisturising topical preparation within the seven days prior to study entry
9. Patients who participated in a study within the three months prior to study entry
10. Patients who are not affiliated to health insurance
11. Patients who are not able or willing to follow the study instructions -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

REFERENCES:
- [Derived] Szepietowski JC, Kemeny L, Mettang T, Arenberger P. Long-Term Efficacy and Tolerability of an Emollient Containing Glycerol and Paraffin for Moderate-to-Severe Uremic Xerosis: A Randomized Phase 3 Study. Dermatol Ther (Heidelb). 2024 Nov;14(11):3033-3046. doi: 10.1007/s13555-024-01287-w. Epub 2024 Oct 18. PMID 39422853

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 237 enrolled patients: one patient not randomized. Among the 118 patients randomized into the V0034CR01B arm, one patient not treated. As such, among the 237 enrolled patients, 235 were treated, ie received test product at least once
Groups:
- V0034CR01B: cream
  V0034CR01B
- V0034 CR 01B Vehicle: cream
  V0034CR01B vehicle
Period: Overall Study
Arm/Group | V0034CR01B | V0034 CR 01B Vehicle
Started | 118 | 118 (Among those 118 patients randomized into V0034 CR 01B vehicle arm, one patient not treated.)
Treated Patients | 118 | 117 (Patients who received test product at least once)
Completed | 88 | 102
Not Completed | 30 | 16

BASELINE CHARACTERISTICS:
Population: 1 patient not randomised
  1 patient in V0034 CR 01B vehicle group not treated
Groups:
- Total: Total of all reporting groups
Arm/Group | V0034CR01B | V0034 CR 01B Vehicle | Total
Number analyzed (Participants) | 118 | 117 | 235
Age, Continuous [Mean (Full Range); unit: years] | 64.8 [26 to 89] | 64.5 [23 to 82] | 64.65 [23 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 53 | 101
  Male | 70 | 64 | 134

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response of Xerosis
Description: Treatment response rate of uremic xerosis on 5 test areas (right lower leg, left lower leg, forearm having no arterio-venous shunt, chest, dorsum of the neck), using a defined 5-point severity scale:
  0 = smooth skin
  1. = patches of fine, powdery scales
  2. = diffuse ashy appearance with many fine scales
  3. = moderate scaling with beginning cracks
  4. = intense scaling, moderate cracks Treatment response was defined as a score of 0 or 1 on all test areas at the end of Period I, and a reduction of at least 2 grades on at least one test area (primary efficacy parameter, Period I).
Time Frame: 28 days
Population: One patient in V0034 CR 01B Vehicle arm randomized but not treated
Measure: Number; unit: participants
Arm/Group | V0034CR01B | V0034 CR 01B Vehicle
Number analyzed (Participants) | 118 | 117
participants | 71 | 48

2. Secondary Outcome: Local Tolerance of V0034 CR 01B After Long-term Use and Patient's Benefit and Acceptability of V0034 CR 01B
Description: At the end of treatment (day 133), patients assessed their overall agreement on the local tolerance of the test product, using a 4-point scale, as follows :
  1. = very satisfactory
  2. = satisfactory
  3. = poorly satisfactory
  4. = not satisfactory at all
Time Frame: 133 days
Measure: Number; unit: participants
Groups:
- V0034CR01B: cream
  V0034CR01B for 28 days (Period I), then treatment free-follow-up (up for 21 days if non persisting lesion and non relapsing lesions (Period II)), then V0034CR01B for 84 days (Period III)
- V0034 CR 01B Vehicle: cream
  V0034CR01B vehicle for 28 days (Period I), then treatment free-follow-up (up for 21 days if non persisting lesion and non relapsing lesions (Period II)), then V0034CR01B for 84 days (Period III)
Arm/Group | V0034CR01B | V0034 CR 01B Vehicle
Number analyzed (Participants) | 118 | 117
participants
  Very satistactory | 68 | 77
  Satisfactory | 26 | 32
  Poorly satisfactory | 5 | 4
  Not satisfactory at all | 6 | 1
  No answer | 13 | 3

ADVERSE EVENTS:
Description: Among the 118 patients randomized into the V0034CR01B arm, one patient not treated.
Arm/Group | V0034CR01B | V0034 CR 01B Vehicle
Serious Adverse Events (participants affected / at risk) | 16/118 | 19/117
Other Adverse Events (participants affected / at risk) | 40/118 | 39/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V0034CR01B (N=118) | V0034 CR 01B Vehicle (N=117)
Death (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Dialysis device complication (Injury, poisoning and procedural complications) | 1 | 0
fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt Thrombosis (Injury, poisoning and procedural complications) | 1 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Disseminated large cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Catheter removal (Surgical and medical procedures) | 1 | 0
Parathyroidectomy (Surgical and medical procedures) | 1 | 0
Renal transplant (Surgical and medical procedures) | 4 | 1
Aortic rupture (Vascular disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 3
Necrosis (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Arteriovenous fistula anevrysm (Injury, poisoning and procedural complications) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Evidence based treatment (Surgical and medical procedures) | 0 | 4
Hospitalisation (Surgical and medical procedures) | 0 | 5
Therapeutic procedure (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V0034CR01B (N=118) | V0034 CR 01B Vehicle (N=117)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Application site erythema (General disorders) | 0 | 1
Application site irritation (General disorders) | 1 | 3
Application site pruritus (General disorders) | 1 | 2
Application site reaction (General disorders) | 1 | 0
Application site vesicles (General disorders) | 2 | 1
Arteriovenous fistule operation (Surgical and medical procedures) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Bacillus infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Blood pressure increased (Investigations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Catheter site infection (Infections and infestations) | 2 | 3
Catheter site pruritus (General disorders) | 1 | 0
catheter site related reaction (General disorders) | 2 | 0
Clavicule fracture (Injury, poisoning and procedural complications) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Eye infection (Infections and infestations) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Haemodialysis-induces symptom (Injury, poisoning and procedural complications) | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Nail infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Paronychia (Infections and infestations) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary track infection (Infections and infestations) | 1 | 4
Vomiting (Gastrointestinal disorders) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Mutual agreement